CLINICAL TRIAL: NCT05612685
Title: Healthcare Providers as Trusted Messengers to Increase Receipt of Tax Credits Among Low-income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kristen R. Choi, PhD, RN, FAAN, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-001575
Record Dates: First submitted 2022-10-20; First posted 2022-11-10 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression; Child Development; Stress; Physical Illness; Health Care Utilization
MeSH Terms: conditions — Depression; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This arm will receive a healthcare provider referral to a tax filing app
  Interventions: Behavioral: Healthcare provider referral to a tax filing app

INTERVENTIONS:
Behavioral: Healthcare provider referral to a tax filing app — Healthcare providers offer a referral to a tax filing app and briefly describe the potential benefits of tax credit receipt

SUMMARY:
The purpose of this study is to pilot test the feasibility and preliminary efficacy of healthcare provider referrals to a tax filing app within parent-child health programs to test whether such referrals can increase receipt of tax credits among low-income parents. The study will use a single-group, pre/post test design with a sample of parents who have a child under 6 years of age. Participants will be recruited from parental-child health programs and clinics in Los Angeles and will complete surveys at baseline, immediately after tax filing season, and six months after tax filing season to assess 1) frequency of tax filing after referral (Feasibility), and 2) pre/posttest changes to parent and child health (preliminary efficacy).

DETAILED DESCRIPTION:
Aims: The purpose of this study is to pilot test the feasibility and preliminary efficacy of healthcare provider referrals to a tax filing app within parental-child health programs whether such referrals can increase receipt of tax credits among low-income parents. The study will use a single-group, pre/posttest design. The primary outcome is feasibility, defined as whether or not participants filed taxes after referral. Secondary outcomes are acceptability of the app and preliminary efficacy of the app on improved parent and child health. Specific aims are to:

1. assess frequency of tax filing among parents referred to a tax filing app (Primary outcome/Feasibility)
2. explore pre/posttest changes to parent and child health after referral (Secondary outcome/Preliminary efficacy).

Design: This pilot study will use a single-group, pre/post-test design to assess the feasibility and preliminary efficacy of healthcare provider referrals to a tax filing app.

Intervention: Referrals to a tax filing app

Setting: The setting for this study is maternal/child health programs and clinics in Los Angeles.

Sample: The target population is parents making less than $75,000 per year in income . Parents will be eligible to participate in the study if they are within the income threshold, have one or more children under six years of age, speak English or Spanish, have access to an internet-enabled device (smart phone or tablet), and have a valid tax filing ID (SSN or ITIN). Parents will be ineligible if they have already filed taxes during the study period or are experiencing an acute mental health crisis (e.g., suicidality). We focus on children under six years of age because this is a critical and sensitive developmental window when interventions have potential for outsized impact on child health.

Procedures: Parents will be recruited during program visits/encounters early in tax season in 2023. Those that provide informed consent to participate in the study will complete a baseline survey and receive the assigned intervention (referral to a tax filing app) the same day or within the same week of their program visit. Parents will complete a follow-up survey to assess outcome measures after they receive tax refunds. A second follow-up survey will be sent 3-6 months later (depending on time of filing, and average time of receipt of tax credit this season) to assess medium-term outcomes.

Outcomes. We will assess the following outcomes. The primary study outcome is feasibility; acceptability and preliminary health efficacy are secondary outcomes.

Feasibility: Self-reported tax filing (items developed for this study) Preliminary efficacy: We will assess pre/posttest changes in the following health-related measures as indicators of preliminary efficacy: 1a) parent overall health rating (PROMIS® Scale v1.2 - Global Health [Hays et al., 2009]; Patient Health Questionnaire- 2 [Kroenke et al., 2003); and 1b) child overall health and developing rating (PROMIS® Early Childhood Parent Report Global Health [Forrest et al., 2014]).

Demographic and family health background information (see survey: age, gender, race/ethnicity, income, social determinants of health, health background, other tax filing characteristics) will be collected to identify characteristics of the sample. In future studies, we intend to study in greater depth the physical health outcomes that might be sensitive to this intervention with longer-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Income <$75,000 per year
* One or more children under 6 years of age
* Has a valid tax filing ID (SSN or ITIN)
* Has access to an internet-enabled device

Exclusion Criteria:

* Experiencing an acute mental health crisis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The target population was parents making less than $75,000 per year seeking maternal/parental or child health services. Parents were eligible to participate in the project if they were within the income threshold, had one or more children under six years of age, spoke English or Spanish, and had a valid tax filing ID (SSN or ITIN). Parents were ineligible if they had already filed taxes or were experiencing an acute mental health crisis (e.g., suicidality).
Period: Overall Study
Arm/Group | Intervention
Started | 21
Completed | 18
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Rate of Tax Filing at 3 Months: Did You File Taxes This Year? YES/NO
Description: Self-reported tax filing status for the current year
Time Frame: 3 months
Population: Participants who completed the follow up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
Participants | 8

2. Primary Outcome: Rate of Tax Filing at 9 Months: Did You File Taxes This Year? YES/NO
Description: Self-reported tax filing status for the current year
Time Frame: 9 months
Population: Individuals who completed the final follow up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
Participants | 8

3. Secondary Outcome: Number of Parents With Positive Depression Score at Baseline
Description: Number of parents with a depression score above the cutoff range (i.e., scores of 3 or greater) on the Patient Health Questionnaire- 2 (score range 0-6, higher scores indicate worse depression symptoms)
Time Frame: Baseline
Population: Baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 18
Participants | 8

4. Secondary Outcome: Number of Parents With Positive Depression Score at 9 Months
Description: as for outcome 3
Time Frame: 9 months
Population: Individuals who completed the follow up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 8
Participants | 1

5. Secondary Outcome: Number of Children With Excellent or Very Good Responses Ratings on Child Development at 9 Months
Description: Number of children with ratings of Excellent or Very Good Responses on child development item in the PROMIS Early Childhood Parent Report Global Health 8a ("How well is your child meeting developmental milestones?" Response options of Excellent, Very Good, Good, Fair, or Poor)
Time Frame: 9 months
Population: Individuals who completed the follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 8
Participants | 6

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
As a single-group feasibility pilot with a small sample, this study cannot establish causal relationships or attribute patterns of findings to the intervention alone. There may have been temporal trends in health or social determinant of health risk related to non-study factors, such as ongoing effects of the coronavirus pandemic or natural disasters in California. We experienced participant attrition and the study inclusion criteria required for tax filing excluded potential participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT05612685/Prot_SAP_ICF_000.pdf